CLINICAL TRIAL: NCT03532425
Title: Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Switching From Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate to Bictegravir/ Emtricitabine/Tenofovir Alafenamide in HIV-1 Infected Virologically Suppressed Adults
Brief Title: B/F/TAF vs Atripla Double-Blind Switch Study in HIV-1 Infected Adults
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties enrolling participants
Sponsor: University of Alberta (Other)
Collaborators: Gilead Sciences (Industry); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BFTAF vs Atripla
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Results first posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- B/F/TAF (Experimental): B/F/TAF + Atripla Placebo
  Each pill is taken once daily, (total of 2 tablets) The blinded treatment phase of this study will last for 52 weeks
  Interventions: Drug: B/F/TAF; Drug: Atripla Placebo
- Atripla (Active Comparator): Atripla + B/F/TAF Placebo
  Each pill is taken once daily, (total of 2 tablets) The blinded treatment phase of this study will last for 52 weeks
  Interventions: Drug: Atripla; Drug: B/F/TAF Placebo

INTERVENTIONS:
Drug: B/F/TAF — B/F/TAF (Bictegravir 50mg/ Emtricitabine 200mg/ Tenofovir Alafenamide 25mg) Tablet taken orally once daily
  Other Names: BIKTARVY®
  Arms: B/F/TAF
Drug: Atripla — Atripla (Efavirenz 600mg/ emtricitabine 200 mg/ tenofovir disoproxil 245 mg) Tablet taken orally once daily
  Arms: Atripla
Drug: B/F/TAF Placebo — Tablet taken orally once daily
  Arms: Atripla
Drug: Atripla Placebo — Tablet taken orally once daily
  Arms: B/F/TAF

SUMMARY:
Atripla (ATP: FTC/TDF/EFV) was the first single pill treatment for HIV and was the most prescribed first-line treatment from approximately 2008 to 2013 for people infected with HIV. However, ATP has not been recommended as a "preferred" treatment for HIV since 2015, due to there now being single pill treatments that work better. There are a lot of people who are still taking ATP and it is working for them. However, it has the potential to cause serious side effects (chronic kidney disease and fractures and serious neurological effects). These side effects are caused by components in ATP (namely the TDF and EFV parts). Also, the efavirenz (EFV) component is not compatible for treatment of Hepatitis C (HCV) - which is often also seen in people who have HIV. For these reasons, there is a need to find a better alternative treatment for these people currently being treated with ATP.

DETAILED DESCRIPTION:
B/F/TAF (bictegravir/FTC/TAF) is an investigational single pill drug treatment drug that contains neither TDF nor EFV. This study is looking at whether changing people to this new drug treatment will continue to suppress their HIV and have fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 seropositive
2. Age > 21 years
3. Receiving ATP > 2 years as their only ART, with HIV-1 RNA < 50 copies/mL at screening and all HIV-1 RNA tests < 100 copies/mL in the past 18 months
4. No documented resistance mutations to the components of ATP
5. Any CD4 count, but no active AIDS-defining opportunistic infections or cancers
6. HBsAg+ permitted if plasma HBV DNA is unquantifiable and the patient does not have decompensated liver disease

Exclusion Criteria:

1. Pregnancy, breastfeeding or planned pregnancy in the next 2 years
2. Documented resistance to the components of ATP
3. Active AIDS-defining opportunistic infection or cancer
4. Cancer in past 3 years, except non melanoma skin cancer
5. Active psychotic disease or active depression that may interfere with study participation according investigator discretion
6. Any illness with a life expectancy less than 2 years
7. eGFR < 50 mL/min
8. Urine protein/creatinine > 40 mg/mmoL
9. Patients who the investigator feels are unlikely to commit to the study requirements for any reason
10. Prescription drug therapy for osteoporosis (calcium and/or vitamin D is allowed)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Shafran, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gallant J, Lazzarin A, Mills A, Orkin C, Podzamczer D, Tebas P, Girard PM, Brar I, Daar ES, Wohl D, Rockstroh J, Wei X, Custodio J, White K, Martin H, Cheng A, Quirk E. Bictegravir, emtricitabine, and tenofovir alafenamide versus dolutegravir, abacavir, and lamivudine for initial treatment of HIV-1 infection (GS-US-380-1489): a double-blind, multicentre, phase 3, randomised controlled non-inferiority trial. Lancet. 2017 Nov 4;390(10107):2063-2072. doi: 10.1016/S0140-6736(17)32299-7. Epub 2017 Aug 31. PMID 28867497
- [Background] Sax PE, Pozniak A, Montes ML, Koenig E, DeJesus E, Stellbrink HJ, Antinori A, Workowski K, Slim J, Reynes J, Garner W, Custodio J, White K, SenGupta D, Cheng A, Quirk E. Coformulated bictegravir, emtricitabine, and tenofovir alafenamide versus dolutegravir with emtricitabine and tenofovir alafenamide, for initial treatment of HIV-1 infection (GS-US-380-1490): a randomised, double-blind, multicentre, phase 3, non-inferiority trial. Lancet. 2017 Nov 4;390(10107):2073-2082. doi: 10.1016/S0140-6736(17)32340-1. Epub 2017 Aug 31. PMID 28867499

RESULTS

PARTICIPANT FLOW:
Groups:
- B/F/TAF: B/F/TAF + Atripla Placebo
  Each pill is taken once daily, (total of 2 tablets) The blinded treatment phase of this study will last for 52 weeks
  B/F/TAF: B/F/TAF (Bictegravir 50mg/ Emtricitabine 200mg/ Tenofovir Alafenamide 25mg) Tablet taken orally once daily
  Atripla Placebo: Tablet taken orally once daily
- Atripla: Atripla + B/F/TAF Placebo
  Each pill is taken once daily, (total of 2 tablets) The blinded treatment phase of this study will last for 52 weeks
  Atripla: Atripla (Efavirenz 600mg/ emtricitabine 200 mg/ tenofovir disoproxil 245 mg) Tablet taken orally once daily
  B/F/TAF Placebo: Tablet taken orally once daily
Period: Overall Study
Arm/Group | B/F/TAF | Atripla
Started | 14 | 14
Completed | 14 | 13
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | B/F/TAF | Atripla | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 11 | 11 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 7 | 11
  Black or African American | 8 | 6 | 14
  Hispanic or Latino | 0 | 1 | 1
  Lebanese | 1 | 0 | 1
  Asian | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Urine Albumin/Creatinine Ratio (UACR)
Description: change in urine albumin/creatinine ratio (UACR)
Time Frame: Baseline and week 48
Population: Data was not collected. Study terminated due to difficulties in enrolling participants.
Arm/Group | B/F/TAF | Atripla
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: HIV-1 RNA
Description: Number of participants with HIV-1 RNA < 50 copies/mL
Time Frame: Week 48
Population: Data was not collected. Study terminated due to difficulties in enrolling participants.
Arm/Group | B/F/TAF | Atripla
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Efavirenz (EFV) Symptom Scores
Description: change in EFV symptom scores from Pittsburgh Sleep Quality Questionnaire (PSQI) global score. PSQI is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. The PSQI global score has a possible range of 0-21. Higher scores represent worse sleep quality.
Time Frame: Baseline and week 4
Population: Data was not collected. Study terminated due to difficulties in enrolling participants.
Arm/Group | B/F/TAF | Atripla
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Urine Protein/Creatinine Ratio (UPCR)
Description: change in urine protein/creatinine ratio (UPCR)
Time Frame: Baseline and week 48
Population: Data was not collected. Study terminated due to difficulties in enrolling participants.
Arm/Group | B/F/TAF | Atripla
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: change in estimated glomerular filtration rate (eGFR)
Time Frame: Baseline and week 48
Population: Data was not collected. Study terminated due to difficulties in enrolling participants.
Arm/Group | B/F/TAF | Atripla
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Bone Mineral Density (BMD) at the Hip
Description: change in bone mineral density (BMD) at the hip
Time Frame: Baseline and week 48
Population: Data was not collected. Study terminated due to difficulties in enrolling participants.
Arm/Group | B/F/TAF | Atripla
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Bone Mineral Density (BMD) at the Spine
Description: change in bone mineral density (BMD) at the spine
Time Frame: Baseline and week 48
Population: Data was not collected. Study terminated due to difficulties in enrolling participants.
Arm/Group | B/F/TAF | Atripla
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: CD4 Lymphocyte Counts
Description: change in CD4 lymphocyte counts
Time Frame: Baseline and week 48
Population: Data was not collected. Study terminated due to difficulties in enrolling participants.
Arm/Group | B/F/TAF | Atripla
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Serum Lipids
Description: change in serum lipids
Time Frame: Baseline and week 48
Population: Data was not collected. Study terminated due to difficulties in enrolling participants.
Arm/Group | B/F/TAF | Atripla
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Adverse Events
Description: number of adverse events
Time Frame: Baseline, week 4, week 12, week 24, week 36, and week 48
Population: Data was not collected. Study terminated due to difficulties in enrolling participants.
Arm/Group | B/F/TAF | Atripla
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout study period of 52 weeks.
Arm/Group | B/F/TAF | Atripla
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/14
Other Adverse Events (participants affected / at risk) | 8/14 | 5/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF (N=14) | Atripla (N=14)
Klebsiella liver abscess (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF (N=14) | Atripla (N=14)
Nausea (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
Back and/or knee pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Common cold/viral respiratory illness (Infections and infestations) | 1 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hemorrhoidectomy (Surgical and medical procedures) | 1 | 0
Elevated ALT (Hepatobiliary disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Total ankle arthroplasty (Surgical and medical procedures) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT03532425/Prot_002.pdf
  • Informed Consent Form (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/25/NCT03532425/ICF_001.pdf